CLINICAL TRIAL: NCT01454713
Title: Retrospective Analysis of Veritas in Breast Reconstruction (RAVE)
Brief Title: Retrospective Analysis of Veritas in Breast Reconstruction
Acronym: RAVE
Status: Completed | Type: Observational
Sponsor: Baxter Healthcare Corporation (Industry)
Collaborators: Synovis Surgical Innovations (Industry)
Responsible Party: Sponsor
Other Study IDs: 10-001
Record Dates: First submitted 2011-10-17; First posted 2011-10-19 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Seroma; Necrosis; Infection
MeSH Terms: conditions — Seroma; Necrosis; Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Veritas: Breast reconstruction with Veritas

SUMMARY:
Retrospective data collection of the use of Veritas in breast reconstruction surgery

DETAILED DESCRIPTION:
This is a multi-center study to retrospectively collect data on the use of Veritas Collagen Matrix in breast reconstruction. Data will be collected on post-operative complications in immediate breast reconstruction and then be compared to literature reported post-operative complication rates associated with the use of acellular dermal matrix in immediate breast reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Patients who underwent mastectomy with immediate breast reconstruction using Veritas collagen matrix
* Patients who underwent mastectomy with single stage procedures or two-stage procedures using Veritas collagen matrix

Exclusion Criteria:

* Patients who underwent delayed breast reconstruction
* Reconstruction with something other than Veritas collagen matrix
* Breasts that were created with DIEP or TRAM procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients who have undergone single-stage or two-stage breast reconstruction surgery with Veritas
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2010-10; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark M Mofid, MD, Principal Investigator — UCSD
Locations (3):
- United States (3):
  - Mark M. Mofid, MD, San Diego, California
  - Michael Meininger, MD, Troy, Michigan
  - Martin Lacey, MD, Saint Paul, Minnesota